CLINICAL TRIAL: NCT05587660
Title: Early Functional Outcomes in Unisplaced Neck of Femur Fracture Treated With Partially Threaded and Fully Threaded Cannulated Screw Fixation in Patients of Age 60 and Above
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Rashida Parveen, Consultant Gynecologist, Nishtar Medical University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NishtarMU123
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Neck of Femur Fracture
Keywords: Cannulated screw; fracture; Hip Harris score
MeSH Terms: conditions — Femoral Neck Fractures; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Randomization to be done through lottery method and then the allocation to be made in both study groups.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partially threaded cannulated screw fixation (Experimental): In Group-A patients, cannulated screw fixation was done using partially threaded screws. In this procedure, first step was insertion of three guide wires under image. The 1st guide wire was inserted immediately above calcar and into femoral head. The second wire was placed posteriorly adjacent to posterior cortex of neck on lateral view. Finally, third guide wire was placed anteriorly and superiorly. Drilling of lateral cortex was done before insertion of screws. Then partially threaded screw fixation was done before removal of guide wires using washers.
  Interventions: Procedure: Fully threaded cannulated screws
- Fully threaded cannulated screws fixation (Experimental): The surgical approach in fully thread cannulated screws fixation group will remain same but instead of partially threaded screwsm fully threaded screws to be used in this group.
  Interventions: Procedure: Fully threaded cannulated screws

INTERVENTIONS:
Procedure: Fully threaded cannulated screws — The most popular method in undisplaced neck of femur fracture include internal fixation by cannulated screws in which screws can be inserted relatively simply and atraumatically as compared to other methods. Screws can be used partially threaded or fully threaded; however studies on fully threaded screw fixation method are inconclusive.

SUMMARY:
This study is done to compare the partially threaded versus fully threaded cannulated screw fixation methods in stable neck of femur fracture in terms of early functional outcomes in patients of age 60 and above. A total of 82 (41 in each group) patients of both genders, aged 60 or above. The Radiographic Union Scale for Hip (RUSH) and Harris Hip score to be used to evaluate fracture healing.

DETAILED DESCRIPTION:
This study is done to compare the partially threaded versus fully threaded cannulated screw fixation methods in stable neck of femur fracture in terms of early functional outcomes in patients of age 60 and above. This is a randomized controlled trial where a total of 82 (41 in each group) patients of both genders, aged 60 or above. All these patients had garden type I or II and were mobile before femoral neck fracture were included. In Group-A patients cannulated screw fixation was done using partially threaded screws and in Group-B patients were treated with fully threaded screws were used. Patients were treated according to following schedule and were followed up at 6 weeks, 3 months and 6 months interval. The Radiographic Union Scale for Hip (RUSH) and Harris Hip score were used to evaluate fracture healing.

ELIGIBILITY:
Inclusion Criteria:

* Patients of garden type I or II fractures.
* All patients to be mobile before femoral neck fracture.

Exclusion Criteria:

* Patients having open fracture.
* Patients with present or past history of chronic kidney disorder.
* Patients presenting with hemorrhage.
* Patient with nervous stroke
* Patients unwilling to be part of this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score (RUSH SCORE) | 6-months
  Harris Hip Score (RUSH SCORE) is the method to assess the result of hip surgery and is intended to evaluate various hip disabilities and methods of treatment. RUSH Score was calculated with "Rradiographic Union Score for Hip (RUSH)", designed to improve intra-and inter-observer reliability when describing the radiographic healing.

CONTACTS AND LOCATIONS:
Locations (1):
- Nishtar Medical University Hospital, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Awais MZ, Salik E, Bokhari SHR, Iqbal MT. A comparative study of early functional outcomes in undisplaced neck of femur fracture treated with partially threaded and fully threaded cannulated screw fixation in patients above 60 years age. Pak J Med Sci. 2023 Sep-Oct;39(5):1531-1534. doi: 10.12669/pjms.39.5.7330. PMID 37680815